CLINICAL TRIAL: NCT06539611
Title: Prospective Cohort Study of a Population at Risk of Psychotic Transition
Acronym: EPEDIP
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Dr Mirvat HAMDAN-DUMONT, Principal investigator, Centre Hospitalier Esquirol
Other Study IDs: 2024-A00720-47
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: At-risk Mental States
Keywords: at-risk mental states; early intervention; psychotic transition; subjective cognitive complaint
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 66 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — This study is observationnal: Questionnaires to assess the endpoint

SUMMARY:
In psychiatry, insight is the patient's awareness of his or her disorder or symptom. Lack of insight also seems to be associated with the presence of anxiety-depressive symptoms.

There are several forms of insight:

* clinical" insight, which is the perception of suffering from a given pathology or symptoms
* cognitive insight (CI), which is the ability to analyse or judge one's own thoughts, beliefs and judgements
* and the insight of cognitive disorders or the subjective perception of the cognitive alterations (or cognitive symptoms) presented. In this study, the investigators will refer to this dimension as 'subjective cognitive complaint' (SCP), in order to differentiate it from cognitive insight, the name of which may lead to confusion.

In schizophrenic disorders, there is a positive correlation between the subjective cognitive complaint SCC, and certain alterations in the neurocognitive assessment, including the attentional dimension. There are scales for collecting SCC in psychotic disorders, such as the SSTICS. To date, there is no scale validated specifically for the UHR population. Thus, the scales used (STICSS, SCoRS, etc.) are validated in populations presenting a characterised psychotic state. Objective impairment is measured during a neurocognitive assessment carried out by a specialised professional: a clinical psychologist specialised in neuropsychology. The cognitive performance of UHR patients is impaired, particularly in terms of cognitive flexibility and self-perception of cognitive disorders, and there may be a discrepancy between the complaint, the objective disorders and their identification as "disorders" by the patient.

Despite this discrepancy, to the investigators knowledge no study to date has investigated a possible link between SCC and psychotic transition in this population. Thus, it is not known whether social class may be a factor in exposure to transition, or whether there is a link at all between social class and risk of transition. The aim of this study is to determine psychotic transition in UHR in a 30 months follow-up, and to determine whether there is a link between SCC and transition.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ;
* Be aged between 15 and 30 ;
* Being assessed by the eDIP (early intervention team "équipe de détection et d'intervention précoce") ;
* Sufficient level of French to understand and express yourself orally and in writing;
* For adults:

Patients who have received informed information about the study and who have signed a consent to participate in the study;

- For minors: Patient who has received informed information about the study and who has signed, as well as the holders of parental authority the minor's consent to participate in the study.

Exclusion Criteria:

* Have already presented a First Psychotic Episode;
* Previous diagnosis of schizophrenia, psychotic disorder or bipolar disorder;
* Being on antipsychotic treatment at the time of inclusion ;
* Known intellectual disability ;
* Pregnant or breast-feeding woman;
* Minors and adults under legal protection.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All youth help-seekers assessed by early intervention team meeting the inclusion criteria will be asked to participate to the study.
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Percent of Psychotic transition in UHR | 30 months
  Use of the CAARMS scale The section on positive symptoms uses a score of symptom intensity (out of 6 points) and frequency (out of 6 points) to determine whether the patient has reached a threshold of mild psychosis (UHR)

SECONDARY OUTCOMES:
Assessment of complaints versus absence of complaints in UHRs | 3 months
  Subjective Cognitive Complaint scale score in UHR within 3 months of assessment. The scale is called SSTICS Subjective Scale to Investigate Cognition in Schizphrenia. Minimal score: 0. Maximal score: 84. Higher scores are related to worse outcomes.
Assessment of attentional impairment versus absence of attentional impairment in UHRs with cognitive complaint | 3 months
  Score at d2R test in the UHR population. d2-R test of attention is a neuropsychological measure of selective and sustained attention and visual scanning speed. The test is computerized. Three main variables are computed and the reported as norm-referenced scores: concentration performance, processed targets and accuracy. Three other variables have only their raw scores reported: errors of omission, errors of commission and errors of commission of "letter" type. Standardized scores consider a test taker's performance in the context of a suitable reference group. The reference group used in this study will be "european population, male and female, 18 - 55 years". The taker's score is plotted as a red line in a graph representing the reference group's performances. Score below 35 is significantly below average. Score over 65 is significantly above average. A higher score is associated with a better outcome.
Date of psychotic transition in UHR patients | 30 months
  The date of transition will be evaluated based on the CAARMS subscale score between follow-up visits.
  The CAARMS Comprehensive Assessment of At-Risk Mental States is a semi-structured assessment tool. The positive symptoms scale is graduated 1 to 6. A higher score is associated with more intense and frequent psychotic symptoms, meaning a worse outcome.
Clinical factors associated with transition in UHR: insight scale BCIS | at baseline: day 1
  Score of Beck Cognitive Insight Scale
  The beck cognitive insight scale is a 15-item self-report consisting of 2 subscales: self- reflectiveness and self-certainty. Overall, cognitive insight is calculated using a composite index, with higher self-reflectiveness relative to self-certainty being indicative of greater cognitive-insight. Composite index scores of three or lower represent low cognitive insight, and ten or above represent good cognitive insight (better outcome).
Clinical factors associated with transition in UHR: self -esteem. | at baseline: day 1
  Score of Rosenberg self-esteem scale
  The Rosenberg self-esteem scale ranges from 0 to 30. Scores below 15 suggest low self-esteem. Scores between 15 and 25 are within normal range (better outcome).
Clinical factors associated with transition in UHR: depression | at baseline: day 1
  Score of Hamilton Depression Scale
  Hamilton depression rating scale ranges from 0 to 54. Score 10- 13 mild depression, 14 to 17 mild to moderate, > 17 moderate to severe depression. Higher score means a worse outcome.
Difference between three groups (NoP no psychosis, UHR and FEP first episode psychosis): insight scale | at baseline: day 1
  Score of Beck Cognitive Insight Scale
  The beck cognitive insight scale is a 15-item self-report consisting of 2 subscales: self- reflectiveness and self-certainty. Overall, cognitive insight is calculated using a composite index, with higher self-reflectiveness relative to self-certainty being indicative of greater cognitive-insight. Composite index scores of three or lower represent low cognitive insight, and ten or above represent good cognitive insight (better outcome).
Difference between three groups (NoP, UHR and FEP): self-esteem. | at baseline: day 1
  Score of Rosenberg self-esteem scale
  The Rosenberg self-esteem scale ranges from 0 to 30. Scores below 15 suggest low self-esteem. Scores between 15 and 25 are within normal range (better outcome).
Difference between three groups ((NoP, UHR and FEP): depression. | at baseline: day 1
  Score of Hamilton Depression Scale Hamilton depression rating scale ranges from 0 to 54. Score 10- 13 mild depression, 14 to 17 mild to moderate, > 17 moderate to severe depression. Higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mirvat B HAMDAN-DUMONT, MD, Principal Investigator — Hospital Esquirol Center
Locations (1):
- Mirvat B HAMDAN-DUMONT, Limoges, France

IPD SHARING:
Plan to Share IPD: Undecided